CLINICAL TRIAL: NCT04247568
Title: The Use of Audiotaped Hypnosis in Promoting Weight Loss Using the Transtheoretical Model of Change
Brief Title: Hypnosis and States of Change to Promote Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Jumana Antoun, Associate Professor of Clinical Family Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBS-2019-0220
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Weight Loss
Keywords: Weight loss; Hypnosis; Adults; Behavior change
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental)
  Interventions: Other: Listening to an audiotape
- Control (Placebo Comparator)
  Interventions: Other: Listening to an audiotape

INTERVENTIONS:
Other: Listening to an audiotape — The participants listen to a audiofile that consists of hypnosis

SUMMARY:
Complementary and alternative therapies for weight loss treatment may be effective. There are few studies showing promise of the use of hypnosis in weight-reduction programs; however, there are lots of bias and more rigorous rials are needed to establish the relationship between hypnosis and weight management. Furthermore, the effect of hypnosis may not be directly related to weight loss but rather on behavioral change. On the basis of the trans theoretical model of change, we hypothesized that audio taped hypnosis would facilitate greater movement through the stages of change toward weight loss as compared to general advice.

OBJECTIVE: The primary aim of this study is to assess the ability of audio taped hypnosis to promote weight loss through its effect on the stages and the processes of change as defined by the Trans theoretical Model of change.

DESIGN: Randomized controlled trial. SETTING: American University of Beirut Medical Center. PARTICIPANTS: Adults with overweight and obesity will be recruited if they had previous attempt to lose weight, are planning to lose weight within the next 6 months or are not satisfied with the results of their current weight loss plan.

INTERVENTIONS: This research will be triple blinded randomized placebo controlled trial. The intervention group will be listening to a hypnotic audio-file on a USB and the control group will be listening to a placebo audio-file on a USB . The hypnotic audio-file will consist of a 20 minutes recording prepared by an experienced hypnotist and the control audio-file will consist of a 20 minutes recording with direct messages targeting lifestyle modification. Follow up visits will take place at 21 days, 3 months, 6 months and 12 months following the intervention to assess for any change in participant's readiness to lose weight.

MAIN OUTCOME MEASURES: The primary outcome will be the difference between the groups in acquiring at least one stage change (upward) as defined by the S-weight from baseline to 3 weeks, 6 months and 12 months post intervention. The secondary outcomes include difference in the mean score of any item of the processes of change between hypnosis audio-file and control audio-file, weight in kg at 3 weeks, 6 and 12 months as compared to baseline weight, decrease in waist circumference in cm as compared to baseline at 6 and 12 months between the hypnosis and control groups, exploring factors that may affect any of the primary and secondary outcomes such as gender, age, educational status, baseline BMI, PHQ2.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 kg/m2 and above, aged 18 to 64 years, able to give written informed consent, fluent in English, all men and women not planning on getting pregnant within the next 12 months, with previous attempts to lose weight, planning to lose weight within the next 6 months or not satisfied with the results of their current weight loss plan.

Exclusion Criteria:

* individuals diagnosed with a psychotic disorder, currently on an antipsychotic medication, pregnant women, women planning on getting pregnant during the study period, not planning on losing weight within the next 6 months, not meeting the inclusion criteria or those who are satisfied with their weight loss progress, and illiterate.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Acquiring at least one stage change (upward) as defined by the S-weight | 21 days, 3 months, 6 months and 12 months
  the difference between the groups in acquiring at least one stage change (upward) as defined by the S-weight from baseline to 3 weeks, 6 months and 12 months post intervention.

SECONDARY OUTCOMES:
Weight change | 21 days, 3 months, 6 months and 12 months
  difference in the weight between hypnosis audio-file and control audio-file, at 3 weeks, 6 and 12 months as compared to baseline weight
difference in the mean score of any item of the processes of change | 21 days, 3 months, 6 months and 12 months
  difference in the mean score of any item of the processes of change between hypnosis audio-file and control audio-file, weight in kg at 3 weeks, 6 and 12 months as compared to baseline
Change in waist circumference in cm as compared to baseline | 6 and 12 months
  decrease in waist circumference in cm as compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Jumana Antoun, Hamra, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antoun J, El Zouki M, Saadeh M. The use of audio self-hypnosis to promote weight loss using the transtheoretical model of change: a randomized clinical pilot trial. PeerJ. 2022 Dec 14;10:e14422. doi: 10.7717/peerj.14422. eCollection 2022. PMID 36536625